CLINICAL TRIAL: NCT02553304
Title: Molecular Features Underlying Racial Differences in Survival of Taiwanese Chronic Lymphocytic Leukemia Patients
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T1914
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The molecular markers to be tested in this project include (but not limited to) cytogenetic abnormalities by fluorescent-in-situ hybridization (FISH), immunoglobulin heavy chain variable region (IGHV) hypermutation status, gene mutations for Notch1, SF3B1, p53, MyD88, and BIRC3, and the expressions for ZAP70 and stem cell factor (SCF).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in adults in Western countries; it is stratified as a subtype of indolent lymphoid malignancy with a long but slowly progressive nature history. However, the clinical course of CLL actually varies widely. Thus, many clinical and molecular features have been identified for outcome predictions. The accurate predictions of prognosis through those factors help for the decision making on the treatment, i.e. to treat patients of high risk of early progression or poor overall survival (OS) with alternative or investigational therapies, while to avoid unnecessary over-treatment for low-risk patients.

CLL is much less prevalent in Eastern countries; presently, most available data on CLL are derived mainly from Western countries. However, a previous report concerning the epidemiology of CLL in Taiwan revealed a drastic increase in the age-adjusted incidence of CLL, a trend not found in Western countries where the incidence rate of CLL remained steadily stable over time. In addition to this epidemiological difference, a population-based analysis has found the overall outcome of CLL, estimated by relative survivals, is steadily much poorer in Taiwanese patients than in US Caucasians. In another report about the cytogenetic profiles in a small cohort of CLL patients in Taiwan, a novel cytogenetic abnormality was found to correlate with poorer outcomes. These reports suggest the existence of ethnic differences in the disease natures of CLL between the East and the West.

To delineate the possible underlying racial differences, especially in the molecular prognostic profiles that might underlie the outcome disparity between Taiwanese and western CLL patients, a comprehensive surveillance of the molecular profiles for CLL in Taiwan is of importance. In this study, we are going to enroll around 250 CLL patients; their clinical parameters will be recorded, their blood samples will be collected for a panel of molecular and cytogenetic factor studies. The molecular markers to be tested in this project include (but not limited to) cytogenetic abnormalities by fluorescent-in-situ hybridization (FISH), immunoglobulin heavy chain variable region (IGHV) hypermutation status, gene mutations for Notch1, SF3B1, p53, MyD88, and BIRC3, and the expressions for ZAP70 and stem cell factor (SCF). These proposed markers include not only the conventional prognostic markers derived from Western studies, and also some novel explorations from our preliminary results, such as SCF and trisomy 3. Through this study, a comprehensive profile of CLL in Taiwan will be established to identify the characteristics of CLL in Taiwanese patients and to address the underlying factors of ethnic differences in the disease nature and outcomes of this disease.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in adults in Western countries; it is stratified as a subtype of indolent lymphoid malignancy with a long but slowly progressive nature history. However, the clinical course of CLL actually varies widely. Thus, many clinical and molecular features have been identified for outcome predictions. The accurate predictions of prognosis through those factors help for the decision making on the treatment, i.e. to treat patients of high risk of early progression or poor overall survival (OS) with alternative or investigational therapies, while to avoid unnecessary over-treatment for low-risk patients.

CLL is much less prevalent in Eastern countries; presently, most available data on CLL are derived mainly from Western countries. However, a previous report concerning the epidemiology of CLL in Taiwan revealed a drastic increase in the age-adjusted incidence of CLL, a trend not found in Western countries where the incidence rate of CLL remained steadily stable over time. In addition to this epidemiological difference, a population-based analysis has found the overall outcome of CLL, estimated by relative survivals, is steadily much poorer in Taiwanese patients than in US Caucasians. In another report about the cytogenetic profiles in a small cohort of CLL patients in Taiwan, a novel cytogenetic abnormality was found to correlate with poorer outcomes. These reports suggest the existence of ethnic differences in the disease natures of CLL between the East and the West.

To delineate the possible underlying racial differences, especially in the molecular prognostic profiles that might underlie the outcome disparity between Taiwanese and western CLL patients, a comprehensive surveillance of the molecular profiles for CLL in Taiwan is of importance. In this study, we are going to enroll around 250 CLL patients; their clinical parameters will be recorded, their blood samples will be collected for a panel of molecular and cytogenetic factor studies. The molecular markers to be tested in this project include (but not limited to) cytogenetic abnormalities by fluorescent-in-situ hybridization (FISH), immunoglobulin heavy chain variable region (IGHV) hypermutation status, gene mutations for Notch1, SF3B1, p53, MyD88, and BIRC3, and the expressions for ZAP70 and stem cell factor (SCF). These proposed markers include not only the conventional prognostic markers derived from Western studies, and also some novel explorations from our preliminary results, such as SCF and trisomy 3. Through this study, a comprehensive profile of CLL in Taiwan will be established to identify the characteristics of CLL in Taiwanese patients and to address the underlying factors of ethnic differences in the disease nature and outcomes of this disease.

Study milestone dates: Study Start (First Patient First Visit Date): July 2015，Recruitment end (Last Patient First Visit): July 2018.，Study end (Last Patient Last Visit): July 2020

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of CLL, either histologically proven or with immunophenotypical pattern by flowcytometry
2. The diagnosis of CLL was made after 2000; the complete medical history and the laboratory data are available for collections.
3. Age of 20 or older
4. Willing to cooperate with the informed consent procedure and the collections of blood samples and medical history.
5. There are no limitations about organ functions, performance status, pregnancy or breast feeding status, or concomitant diseases or medicines.
6. The patient's peripheral hemogram shows apparent leukocytosis (>15 k/μL) with lymphocytosis (lymphocytes+atypical lymphocytes >55%); the data should me within 3 months before study enrollment.

Exclusion Criteria:

1. The patient's past history, including the diagnostic test results, the prior CLL-related treatment courses, the drug history, et.al, is not available.
2. The patient cannot complete the informed consent procedures.
3. The diagnosis is T-CLL, or the patients have been in complete remission without peripheral leukemia cells.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic lymphocytic leukemia (CLL)Patient
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
molecular prognostic profiles | 2 years
  establish the biological profiles of CLL

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, MD, Study Director — Taiwain Cooperation Organization Group,NHRI,Taiwain